CLINICAL TRIAL: NCT05246475
Title: Simultaneous PET-MRI for Comparison of Advanced DW-MRI Techniques and EF5-PET in the Detection of Hypoxia in Head and Neck Cancer
Brief Title: Measurement of Head and Neck Tumor Hypoxia With PET-MRI
Acronym: EF5NECK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Jussi Hirvonen, Radiologist, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T255/2021
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be scanned with both MRI and PET.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET-MRI (Experimental): Simultaneous 18F-EF5 PET and DW-MRI
  Interventions: Diagnostic Test: PET-MRI

INTERVENTIONS:
Diagnostic Test: PET-MRI — Simultaneous PET-MRI measurement

SUMMARY:
This study is designed to evaluate the performance of advanced magnetic resonance (MR) imaging in the assessment of tumor hypoxia using [18F]EF5 positron emission tomography (PET) as a reference in head and neck cancer patients. Low oxygen level or hypoxia contributes to radiotherapy resistance. Therefore, a clinically applicable method to detect tumor hypoxia is of great importance.

DETAILED DESCRIPTION:
This is a non-randomized prospective study which aims to compare [18F]EF5 PET data and MR imaging data acquired with simultaneous PET/MR imaging. Hypoxic tumor tends to be more aggressive than its non-hypoxic counterpart since hypoxia promotes invasive tumor growth and metastatic spread of the disease. The detrimental effect of hypoxia on outcome of radiotherapy (RT) is especially important in head and neck cancer.

EF5 is a comprehensively studied hypoxia-avid compound, which is utilized in radiolabeled form in [18F]EF5 PET imaging detecting tumor hypoxia. IVIM (intra-voxel incoherent motion) is novel technique based on diffusion-weighted MRI (DWI), which allows for the distinction between tissue perfusion and diffusion without the need for intravenous contrast agent. This study aims to investigate the potential of novel MRI techniques for tumor hypoxia assessment in HNC.

The specific aims of the current study are:

1. To characterize the voxel-level relationship between diffusion characteristics in tumor tissue, as measured with DW-MRI, and tumor hypoxia, as measured with [18F]EF5-PET, leveraging the state-of-the-art simultaneous MRI/PET measurement;
2. To employ IVIM-based modeling of DW-MRI signal using multiple b-values to optimize the diffusion metrics that most closely predict tumor hypoxia, and compare those with the perfusion metrics from DCE;
3. To develop models based on novel radiophenotypic analyses of MRI data (radiomics) and machine learning algorithms to find MRI patterns that best predict tumor hypoxia at the patient sample level.

The only intervention for participating subjects is an additional [18F]EF5-PET/MR scan, which is not used for any clinical purposes. All study subjects will undergo standard diagnostic and treatment procedures according to clinical routine.

A standard dose of about 300 MBq of the radiotracer [18F]EF5 will be administered intravenously via an upper extremity vein. About 180 min after tracer injection, radioactivity will be followed in the neck area with the PET/MRI device for about 20 min. [18F]EF5 uptake will be modeled as standard uptake value (SUV), and tumor-to-background ratios (TBR) will be calculated.

The MRI protocol will include anatomical sequences covering the primary tumor as well as the neck for lymph node metastases. Several DW-MRI methods will also be employed. In total, MRI experiments will be completed in about 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 80 years old
* Sex: male or female
* Language spoken: Finnish or Swedish
* Performance status: Karnofsky score 70 or better or WHO performance status 2 or better
* Mental status: Patients must be able to understand the meaning of the study
* Diagnosis: Histological, cytological and clinical findings are consistent with squamous cell carcinoma of the head and neck (oral cavity, pharynx or larynx)
* Primary tumor diameter as determined clinically or from contrast enhanced CT or MRI scan must be at least 20 mm
* Patients with nodal neck metastases of head and neck cancer are eligible
* Informed consent: The patient must sign the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff
* Gravidity: Patient, if female, must not be pregnant or lactating at the time of the study

Exclusion Criteria:

* Any previously known contraindication of MR Imaging (including but not limited to metallic implants or foreign bodies, pacemakers or other cardiac implantable electronic devices, MR-incompatible prosthetic heart valves, contrast allergy, claustrophobia)
* Prior Medical History: Patient must have no history of serious haematologic, cardiovascular, liver or kidney disease. Since none of these is an absolute contraindication for inclusion final judgement will be left to the investigators.
* Prior Therapy: Patient must have no history of previous chemotherapy, biological therapy, immunotherapy, radiotherapy or major surgery for treatment of head and neck cancer
* Infections: Patient must not have an uncontrolled serious infection
* Advanced disease: Patient is not eligible for curative cancer treatment due to advanced disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
PET-MRI correlation | 1 day
  Voxel level correlation of DW-MRI and PET estimates

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Hirvonen, MD, PhD, Principal Investigator — Radiologist
Locations (1):
- Turku University Hospital, Turku, G102881, Finland

IPD SHARING:
Plan to Share IPD: No